CLINICAL TRIAL: NCT00726752
Title: A Phase 1 Study In Patients With Advanced Solid Tumor To Evaluate The Pharmacokinetics And Safety Of AG-013736 At Single Doses Of 5 mg, 7 mg And 10 mg, And At Multiple Doses
Brief Title: A Study In Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061044
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Neoplasms
Keywords: solid tumor; Axitinib; Pharmacokinetics; Phase 1
MeSH Terms: conditions — Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib (Experimental)
  Interventions: Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Axitinib (AG-013736) — Three single dose level of AG-013736 (5 mg, 7 mg and 10 mg) will be given for all patient. After single dosing at each dose level, multiple doses of 5 mg twice a day (BID) will be started.

SUMMARY:
This study designed to evaluate the pharmacokinetics and safety of AG-013736 at single doses and multiple doses

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically or cytologically diagnosed with advanced solid tumors
* Patients for whom standard therapies have not been effective, or for whom there are no suitable therapies
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1 or 2
* Patients with no uncontrolled hypertension

Exclusion Criteria:

* Patients who have central lung lesions involving major blood vessels
* Patients who require anticoagulant therapy.
* Patients with active epilepsy seizure or symptoms, with brain metastases requiring treatment, with spinal cord compression and with carcinomatous meningitis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Kobe, Hyōgo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061044&StudyName=A%20Study%20In%20Patients%20With%20Advanced%20Solid%20Tumor

RESULTS

PARTICIPANT FLOW:
Groups:
- AG-013736: Single Dosing: Participants received single AG-013736 5 mg, followed by 7 mg, and subsequently 10 mg. After the single dose at each dose level, participants were monitored for at least 48 hours prior to the next dosing. Multiple Dosing (28-day cycle ): After the monitoring period following the 10 mg single dose, participants received multiple doses of AG-013736 at 5 mg twice daily (BID) at approximately 12 hours apart. The treatment was continued until participants experienced intolerable toxicity or progressive disease.
Period: Overall Study
Arm/Group | AG-013736
Started | 6
Completed | 0
Not Completed | 6
Not completed — Lack of Efficacy | 6

BASELINE CHARACTERISTICS:
Arm/Group | AG-013736
Number analyzed (Participants) | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 53.8 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Single Dose: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 24, and 32-hour postdose
Population: Pharmacokinetic analysis set was defined as all enrolled participants who received at least 1 dose of the study medication and who completed pharmacokinetic blood sampling for at least 1 day.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 6
ng/mL
  5 mg Single Dose | 20.732 (14.492)
  7 mg Single Dose | 32.007 (28.223)
  10 mg Single Dose | 53.123 (60.921)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time Infinity (AUCinf)
Description: AUCinf is obtained from AUC (0 - t) plus AUC (t - infinity).
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 24, and 32-hour postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 6
ng*hr/mL
  5 mg Single Dose | 180.25 (154.90)
  7 mg Single Dose | 228.45 (183.12)
  10 mg Single Dose | 379.12 (345.50)

3. Primary Outcome: Single Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 24, and 32-hour postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AG-013736
Number analyzed (Participants) | 6
hours
  5 mg Single Dose | 4.1000 [3.950 to 6.020]
  7 mg Single Dose | 4.0000 [0.983 to 9.880]
  10 mg Single Dose | 4.0150 [2.050 to 6.000]

4. Primary Outcome: Single Dose: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 24, and 32-hour postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AG-013736
Number analyzed (Participants) | 6
hours
  5 mg Single Dose | 4.778 (2.815)
  7 mg Single Dose | 5.088 (2.592)
  10 mg Single Dose | 5.880 (3.456)

5. Secondary Outcome: Multiple Dose: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax at multiple dosing
Time Frame: Cycle 1 Day 15 predose in the morning, and 0.5, 1, 2, 4, 8 and 12 hour postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 6
ng/mL | 25.933 (21.703)

6. Secondary Outcome: Multiple Dose: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: The dosing interval was 12 hours in this study.
Time Frame: Cycle 1 Day 15 predose in the morning, and 0.5, 1, 2, 4, 8 and 12 hour postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 6
ng*h/mL | 164.55 (128.15)

7. Secondary Outcome: Multiple Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax at multiple dosing
Time Frame: Cycle 1 Day 15 predose in the morning, and 0.5, 1, 2, 4, 8 and 12 hour postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AG-013736
Number analyzed (Participants) | 6
hours | 4.0400 [3.930 to 7.700]

8. Secondary Outcome: Multiple Dose: Accumulation Ratio for Cmax (Rac Cmax) and Accumulation Ratio for AUCtau (Rac AUCtau)
Description: Rac Cmax is obtained from Cmax (Cycle 1, Day 15) divided by Cmax (Cycle 1, Day 1) Rac AUCtau is obtained from AUCtau (Cycle 1, Day 15) divided by AUCtau (Cycle 1, Day 1)
Time Frame: Cycle 1 Day 15 predose in the morning, and 0.5, 1, 2, 4, 8 and 12 hour postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AG-013736
Number analyzed (Participants) | 6
ratio
  Rac Cmax | 1.3540 (0.5335)
  Rac AUCtau | 1.4185 (0.3951)

9. Secondary Outcome: Percent Change From Baseline in Soluble Vascular Endothelial Growth Factor Receptor 1, 2, and 3 (s-VEGFR1, s-VEGFR2 and s-VEGFR3), Vascular Endothelial Growth Factor (VEGF), Soluble Stem Cell Factor Receptor (s-KIT )
Description: Percent change from baseline is obtained from (observed value minus baseline value) divided by baseline value multiplied by 100 in each parameter, i.e., s-VEGFR1, VEGFR2, s-VEGFR3, s-KIT, and VEGF
Time Frame: Prior to the initial dose (baseline) and Day 1 of Cycle 2
Population: Pharmacodynamic analysis set was defined as all enrolled participants who received at least 1 dose of the study medication and who completed pharmacodynamic blood sampling for at least 1 day.
Measure: Median (Full Range); unit: percent
Arm/Group | AG-013736
Number analyzed (Participants) | 6
percent
  s-VEGFR1 | -29.15 [-31.4 to -25.3]
  s-VEGFR2 | -33.16 [-58.4 to -26.2]
  s-VEGFR3 | -56.38 [-66.2 to -42.1]
  s-KIT | -14.59 [-23.7 to -5.2]
  VEGF | 179.52 [37.0 to 1444.6]

10. Secondary Outcome: Number of Participants With Best Overall Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progression of Disease (PD) According to the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0)
Description: CR was defined as the disappearance of all target and nontarget lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters (SLD) of the targeted lesions. CR and PR had to be documented on 2 occasions separated by at least 4 weeks. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify as PD being demonstrated during the first 8 weeks. PD was defined as at least a 20% increase in the SLD of target lesions compared to the smallest SLD since the study treatment started.
Time Frame: Up to 470 days
Population: Anti-tumor response analysis set was defined as all participants with at least 1 target lesion according to RECIST and who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | AG-013736
Number analyzed (Participants) | 6
participants
  CR | 0
  PR | 0
  SD | 3
  PD | 3

11. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any adverse events, adverse events graded as Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 Grade 3 or higher , serious adverse events, and adverse events resulted in discontinuation.
Time Frame: Up to 470 days of treatment plus 28-days follow-up
Population: Safety analysis set was defined as all enrolled participants who received the study drug at least once in this study (same as the full analysis set:FAS).
Measure: Number; unit: participants
Arm/Group | AG-013736
Number analyzed (Participants) | 6
participants
  Any adverse events | 6
  Any serious adverse events | 1
  Any Grade-3 or -4 adverse events | 4
  Any Grade-5 adverse events (= death) | 1
  Discontinuation due to adverse events | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | AG-013736
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (N=6)
Disease progression (General disorders) | 1 — Caused death.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (N=6)
Thyroiditis chronic (Endocrine disorders) | 1
Eye irritation (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 5
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Nasopharyngitis (Infections and infestations) | 2
Paronychia (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 3
Blood amylase increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 3
Blood potassium increased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 2
Blood thyroid stimulating hormone increased (Investigations) | 4
Blood urine present (Investigations) | 1
Lipase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Thyroglobulin increased (Investigations) | 1
Thyroxine free decreased (Investigations) | 2
Thyroxine free increased (Investigations) | 1
Tri-iodothyronine free decreased (Investigations) | 2
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 4
Menstruation irregular (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.